CLINICAL TRIAL: NCT03269344
Title: Randomized Phase III, Double-Blind, Placebo Controlled Study of Prophylactic Gabapentin for the Reduction of Radiation Therapy Induced Pain During the Treatment of Oropharyngeal Squamous Cell Carcinoma
Brief Title: Gabapentin for the Reduction of Radiation Therapy Induced Pain During the Treatment of Oropharyngeal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Andrew Cook, Resident Physcian, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HFHS-Gabapentin/RT Study
Record Dates: First submitted 2017-06-05; First posted 2017-08-31 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): Standard supportive care during definitive treatment plus placebo
  Interventions: Drug: Placebo Oral Capsule
- Experimental Arm (Experimental): Gabapentin plus standard supportive care
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin is an anticonvulsant and has been used to manage neuropathic pain and is FDA-approved for the treatment of post-herpetic neuralgia and partial onset seizures
  Arms: Experimental Arm
Drug: Placebo Oral Capsule — Placebo
  Arms: Control Arm

SUMMARY:
Strategies to minimize and mitigate external beam radiation therapy related mucositis and pain during the treatment of head and neck cancer remain limited. The investigators hypothesize that gabapentin could be used to delay or reduce treatment-related pain, reliance on opioid medication, and improve the quality of life for these patients.

DETAILED DESCRIPTION:
The specific aims of this proposed study include the following:

* Evaluate the reduction or delay of mucositis related pain and morbidity with the use of gabapentin in patients with stage III or IV oropharyngeal squamous cell carcinoma undergoing definitive radiation with concurrent chemotherapy as part of their cancer management, compared to standard supportive side effect mitigation - using patient reported quality of life endpoints such as the Patient-Reported Oral Mucositis Symptoms (PROMS) scale.
* Assess morphine-equivalent opioid use in both treatment arms by collecting the patient's narcotic use in the previous 24-hour period at each weekly evaluation during radiation treatment.
* Report on change in Speech and swallow performance, as measured by the Performance Status Scale (PSS) for Head and Neck Cancer Patients
* Evaluate changes in weight from baseline throughout treatment between the two arms.
* Assess feeding tube requirements during treatment.
* Evaluate the adverse events associated with gabapentin.
* Evaluate the severity of radiation mucositis (grade 3-4, CTCAE, v. 4)

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with combination chemotherapy and radiation therapy daily for locally advanced (stage III-IV) squamous cell carcinoma of the oropharynx.
* Age ≥ 18.
* ECOG performance status ≤ 1.
* Patients must provide study specific informed consent prior to study entry and be able to fill out toxicity and quality of life related questionnaires.

Exclusion Criteria:

* Patients may not be receiving gabapentin, any other investigational agents, or other anticonvulsants.
* Patients with metastatic disease are excluded from this clinical trial.
* Patient with allergies or hypersensitivity to gabapentin.
* Patients receiving surgery as part of their definitive management.
* Patients who have received prior chemotherapy or radiation therapy.
* Patients unable to complete the required forms; however, verbal completion is adequate if recorded on the form daily.
* Uncontrolled serious illness including, but not limited to, ongoing or serious active infection requiring IV antibiotics for over 30 days, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzan Siddiqui, MD PhD, Study Chair — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cook A, Modh A, Ali H, Sheqwara J, Chang S, Ghanem T, Momin S, Wu V, Tam S, Money S, Han X, Fakhoury L, Movsas B, Siddiqui F. Randomized Phase 3, Double-Blind, Placebo-Controlled Study of Prophylactic Gabapentin for the Reduction of Oral Mucositis Pain During the Treatment of Oropharyngeal Squamous Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2022 Mar 15;112(4):926-937. doi: 10.1016/j.ijrobp.2021.11.012. Epub 2021 Nov 20. PMID 34808255

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 65 patients were enrolled, 7 more were excluded from analysis, leaving 58 patients analyzed. These patients were excluded because they received immunotherapy (n=1), pursued treatment elsewhere (n=2), developed acute kidney injury (n=1), and refused to take medication during the first two weeks of treatment (n=3).
Period: Overall Study
Arm/Group | Control Arm | Experimental Arm
Started | 33 | 32
Completed | 29 | 29
Not Completed | 4 | 3
Not completed — Protocol Violation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Experimental Arm | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (8.5) | 60.2 (10.4) | 59.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Smoking Status [Count of Participants; unit: Participants] — Stratification variable
  Participants | 7 | 9 | 16
Primary Site [Count of Participants; unit: Participants]
  Oropharynx-base of tongue | 10 | 11 | 21
  Oropharynx-soft palate | 1 | 0 | 1
  Oropharynx-tonsil | 12 | 17 | 29
  Oropharynx-vallecula | 2 | 0 | 2
  Oropharynx-not specified | 3 | 1 | 4
  Unknown primary | 1 | 0 | 1
HPV Status [Count of Participants; unit: Participants]
  Negative | 5 | 3 | 8
  Positive | 23 | 26 | 49
  Unknown | 1 | 0 | 1
Clinical T Stage [Count of Participants; unit: Participants] — Patients were staged according to the American Joint Committee on Cancer staging system 8th edition (2017) for oropharyngeal tumors. Higher numbers indicated higher stage/more advanced tumors.
  Participants
    1 | 8 | 6 | 14
    2 | 11 | 10 | 21
    3 | 5 | 7 | 12
    4 | 2 | 4 | 6
    4a | 1 | 1 | 2
    4b | 1 | 0 | 1
    Tx or T0 | 1 | 1 | 2
Clinical N Stage [Count of Participants; unit: Participants] — Patients were staged according to the American Joint Committee on Cancer staging system 8th edition (2017) for oropharyngeal tumors. Higher numbers indicated higher stage/more advanced tumors.
  Participants
    0 | 0 | 2 | 2
    1 | 17 | 15 | 32
    2 | 7 | 6 | 13
    2a | 0 | 1 | 1
    2b | 3 | 1 | 4
    2c | 2 | 1 | 3
    3 | 0 | 3 | 3
Type of Chemotherapy [Count of Participants; unit: Participants]
  Carboplatin-based | 3 | 4 | 7
  Cisplatin every 3 weeks | 16 | 16 | 32
  Cisplatin weekly | 10 | 9 | 19
Opioid Use at Baseline [Count of Participants; unit: Participants] | 3 | 4 | 7
Gross Tumor Volume of Primary Tumor [Mean (Standard Deviation); unit: cubic centimeter (cc)] | 22.0 (17.2) | 21.5 (18.5) | 21.8 (17.9)
Gross Tumor Volume Total (cc) [Mean (Standard Deviation); unit: cc] | 50.3 (40.8) | 49.2 (31.5) | 49.8 (36.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life From Mucositis-related Pain Measured by the Patient-Reported Oral Mucositis Symptoms (PROMS) Scale From Baseline to Follow-up
Description: Scale tile: Patient Reported Oral Mucositis Symptoms scale, range 0-1000, higher scores indicate worse outcomes
Time Frame: Evaluated change in scores from baseline to 6 weeks post-treatment, approximately 13 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
score on a scale | 20.1 (16.8) | 29.1 (22.5)
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.11, ANOVA

2. Secondary Outcome: Change in Total FACT-HN Scores From Baseline to Follow-up
Description: Scale: Functional Assessment of Cancer Therapy-Trial Outcome (FACT-HN), range 0-148, higher scores indicate better outcomes
Time Frame: Administered at baseline and at 6-week follow-up endpoint, approximately 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
units on a scale | -15.0 [-19.5 to -2.5] | -20.0 [-25.8 to -11.8]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Average Opioid Use, Measured in Morphine Equivalents Per Day.
Time Frame: Over the entire study period from baseline to follow-up, approximately 13 weeks
Measure: Median (Inter-Quartile Range); unit: Daily morphine equivalents
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
Daily morphine equivalents | 15.6 [6.7 to 32.2] | 22.2 [13.3 to 35.0]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in PRO-CTCAE Scores From Baseline to Follow-up
Description: Scale: Patient-reported outcomes of Common Terminology Criteria for Adverse Events (PRO-CTCAE), 5-point Likert scale, higher scores indicate worse outcomes. Range of scores 0-40 (min-max).
Time Frame: Evaluated change in scores from baseline to 6 weeks post-treatment, approximately 13 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
units on a scale | 1.0 [-2.0 to 6.0] | 6.5 [3.5 to 11.8]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percent Weight Lost
Description: Percent weight lost from baseline to week 7 of treatment (end of treatment)
Time Frame: Percent change from baseline to week 7 of treatment
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
Percent change | -10.7 [-14.4 to -7.8] | -11.4 [-15.6 to -8.0]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Feeding Tube Placement
Description: Measure of number of patients who required feeding tube placement at any time during the study period
Time Frame: Evaluated placement of feeding tube from baseline (start of radiation) to 6 weeks post-treatment, approximately 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 29 | 29
Participants | 6 | 18
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p < 0.01, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse effects data were collected from baseline, throughout the 7 week treatment course, and at the 6-week post-treatment follow-up timepoint. Thus, this time period was about 14 weeks.
Arm/Group | Control Arm | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03269344/Prot_SAP_000.pdf